CLINICAL TRIAL: NCT04259775
Title: Guided User-initiated Insulin Dose Enhancements (GUIDE) to Improve Outcomes for Youth With Type 1 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Needed FDA approval
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000027002; 2K12DK094714-06 (NIH)
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
Keywords: automated insulin dose adjustment; continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated Insulin Dose Adjustment (AIDA) (Active Comparator): Using the AIDA system to assist the parents of children with T1D make insulin dose adjustments
  Interventions: Device: Automated Insulin Dose Adjustment
- Control (Active Comparator): Standard Care - change in therapy settings effected a regularly scheduled patients visits
  Interventions: Device: Control

INTERVENTIONS:
Device: Automated Insulin Dose Adjustment — The system originally developed at Boston Children's Hospital, obtains CGM, insulin delivery, and activity data, from the cloud each day at approximately 8:00 PM using an Application Program Interface (API) calls to commercial companies (primarily Glooko and Tidepool) that aggregate data from different devices used to manage glucose levels in individuals. A detailed statistical and control analysis (see preliminary data study 1 for algorithm details) of the data are then conducted to determine if a change in therapy is required. If the analysis indicates a change in therapy is required, the patient or parent is notified by text or email directing then to a web portal detailing the change. The patient or parent can accept or modify the recommended change. If a change is made, the AIDA system confirms that the change is correctly implemented into the patient's pump or Bluetooth enabled pen when the patient next uploads the device data to the cloud.
  Arms: Automated Insulin Dose Adjustment (AIDA)
Device: Control — Standard Care - change in therapy settings effected at regularly scheduled patient visits
  Arms: Control

SUMMARY:
We propose conducting a pilot randomized study to assess the feasibility of using the automated insulin dose adjustment (AIDA) system to assist the parents of children with Type 1 Diabetes to make insulin dose adjustments between visits with their diabetes provider. Study results will be used to inform a larger RCT with an anticipated primary outcome of change in HbA1c in patients managed with either standard care (changes in therapy settings effected at regularly scheduled patients visits) or AIDA guided care.

DETAILED DESCRIPTION:
Screening & End of 3-Week Run-in Period (Visit 1, Week 0) : Screening will be conducted by invitation to potentially eligible subjects. The study will be explained and written informed consent will be obtained from parents or patients (when 18 years of age or older) prior to conducting any study-related procedures. After written informed consent and patient assent (when <18 years of age) have been obtained, potential participants will undergo a history and physical exam. Girls of childbearing potential will have a urine pregnancy test performed at the time of the enrollment visit and the need for contraception for the entire duration of the study will be discussed. At this and all other study visits, participants/parents will meet with a diabetes care provider (i.e., a physician, nurse practitioner, or physician assistant) who will carry out a comprehensive review of diabetes management and review blood glucose and ketone records. The treatment regimen will be adjusted as clinically indicated during the initial screening visit and baseline data (including CGM and insulin dose data) will be collected in all participants during the 3-week run-in period of the study; HbA1c levels will be measured at the end of the 3-week baseline period in all eligible participants.

Baseline data obtained at the screening or 3-week baseline visit will include:

* Demographic characteristics, including family income, highest parental education attained, and number of individuals in the home
* 3-week data regarding CGM, insulin dose and Fitbit data
* Anthropometric measures (height, weight, BMI, vital signs) and physical exam
* Current diabetes care practices (frequency of self-monitored blood glucose (SMBG), insulin dosing, review of blood glucose values)
* Medical History: duration of diabetes, comorbidities, past medical history, social history, family history, medications, and allergies
* Additional diabetes history including current/past use of CGM, insulin pump, and other modes of diabetes technology
* Frequency of Emergency Department visits due to decompensated diabetes (i.e., hyperglycemia, ketosis and DKA) over the past 6 months
* Baseline laboratory assessment including lipid panel and urine microalbumin
* Psychosocial Questionnaires will be administered

  1. Hypoglycemia Fear Survey (parent and child)
  2. Pittsburgh Sleep Quality Index
  3. Diabetes Treatment Satisfaction Questionnaire (DTSQ, DTSQc), which includes eight items, six of which form a scale (scored 0-36) in which higher scores indicate greater treatment satisfaction
  4. Diabetes-specific emotional distress using Problem Areas in Diabetes scale

After collection of all baseline data, eligible participants will be randomized to either the control or intervention group and receive instructions for the study. Participants will also be provided with a FitBit and instructed to wear this for the duration of the study to track activity levels. Participants in the intervention group will be required to upload their diabetes devices to Tidepool each week for the duration of the study. Tidepool is program used at Yale Pediatric Diabetes clinics as the current standard of care for uploading devices (pumps, CGMs, Bluetooth enabled pens) in our clinics and is HIPAA compliant. Participants may contact the Yale Diabetes Team for insulin dose adjustments or the study team at any point during the study if they have a question about the study.

Visit 2 (Week 13) & Visit 3 (Week 26): At these visits, all participants will meet with a diabetes care provider who will carry out a comprehensive review of diabetes management and review blood glucose and insulin records. Diabetes devices will be downloaded, and glycemic trends and insulin dosing regimens will be reviewed. The treatment regimen will be adjusted as clinically indicated.

After 26 weeks in the study, intervention group parents will be asked to participate in focus groups to discuss the study. These meetings will take place at the Yale Pediatric Diabetes Research Center.

ELIGIBILITY:
Inclusion Criteria:

i. Clinical diagnosis of type 1 diabetes for at least 1 year ii. Ages 7-21 years iii. Participants 18 years of age must be able to read and provide written consent iv. Participants under 18 years of age must be able to read and provide written assent v. Participants are managed using an insulin pump or multiple daily injections vi. Participant has a CGM or is willing to wear a CGM for the duration of the study

Exclusion Criteria:

I. Hemoglobin A1c <7.5% or > 10.0% ii. Recent history of more than 1 episode of diabetic ketoacidosis (DKA) in the past 4 months iii. Treatment with glucose lowering drugs other than insulin iv. Females who are pregnant, lactating, or planning to become pregnant in the next 6 months v. Another medical condition that precludes participation in the study.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Percent of patients at target range from baseline to 13 week | 13 weeks
  Based on continuous glucose monitoring. Target range is defined as 70- 180 mg/dL
Percent of patients at target range from baseline to 26 weeks | 26 weeks
  Based on continuous glucose monitoring. Target range is defined as 70- 180 mg/dL

SECONDARY OUTCOMES:
Change from baseline in HbA1c | 13 weeks
  This outcome will determine if there was a change in HbA1c levels from baseline to 13 weeks based on continuous glucose monitoring
Nighttime hypoglycemic defined as the % of time spent <55 mg/dL | Baseline
  Based on continuous glucose monitoring
Nighttime hypoglycemic defined as the % of time spent <55 mg/dL | 13 week
  Based on continuous glucose monitoring
Nighttime hypoglycemic defined as the % of time spent <55 mg/dL | 26 week
  Based on continuous glucose monitoring
Nighttime hypoglycemic defined as the % of time spent under 70 mg/dL | Baseline
  Frequency of nighttime hypoglycemic events
Nighttime hypoglycemic defined as the % of time spent under 70 mg/dL | 13 week
  Frequency of nighttime hypoglycemic events
Nighttime hypoglycemic defined as the % of time spent under 70 mg/dL | 26 week
  Frequency of nighttime hypoglycemic events
Percent of the recommendations that are accepted or modified by the family | 26 week
  Percent of the recommendations that are accepted or modified by the family
Hypoglycemia Fear Survey | 26 weeks
  This will be administered to the child and parent. The survey consists of 23 questions. Questions are answered using a 5 point likert scale ranging from never, rarely, sometimes, often, and always. The administration time is 10 minutes. The higher scores entail greater worry.
Pittsburgh Sleep Quality Survey (PSQI) | 26 weeks
  The survey consists of 10 questions. The Questions relate to usual sleep habits over the last month, including time it takes to fall asleep, usual bedtime, hours of sleep per night, as well as questions about the frequency of sleep issues (not during the past month, less than once per week, once or twice per week, or three or more times per week). Higher scores suggest poorer sleep quality. The administration time is 5 minutes.
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 26 weeks
  This will be administered to the parent and teen. The survey consists of 12-24 questions that are based on a likert scale ranging from 0 to 6. Higher scores entail greater satisfaction. The administration time is 10 minutes.
Problem Areas in Diabetes Scale (PAID) | 26 weeks
  This is a questionnaire with 20 questions scaled from 0 to 4 on a likert scale. Questions involve feelings and emotional distress related to diabetes. Higher scores entail a more serious problem related to diabetes. The Administration time is 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Nally, MD, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No